CLINICAL TRIAL: NCT02815124
Title: Randomized Controlled Trial of Image-Guided Cochlear Implant Programming Versus Standard of Care
Brief Title: Trial of Image-Guided Cochlear Implant Programming Versus Standard of Care
Acronym: IGCIP vs SOC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding secured and staffing changes resulting in no personnel to assist with study tasks.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Robert F. Labadie, Vice Chair, Chief Research Officer, Professor of Otolaryngology-Head and Neck Surgery, Professor of Biomedical Engineering, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160461; R01DC014462 (NIH)
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cochlear Implant
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Cochlear Implant programming using standard of care
  Interventions: Other: Standard of Care
- Image-Guided Cochlear Implant Programming (Experimental): Cochlear Implant programming using Image-Guided Cochlear Implant Programming
  Interventions: Other: Image-Guided Cochlear Implant Programming

INTERVENTIONS:
Other: Standard of Care — Post Cochlear Implant surgery, subject will receive activation/programming of their implant using Standard of Care
  Arms: Standard of Care
Other: Image-Guided Cochlear Implant Programming — Post Cochlear Implant surgery, subject will receive activation/programming of their implant using Image-Guided Cochlear Implant Programming
  Arms: Image-Guided Cochlear Implant Programming

SUMMARY:
Cochlear implants are surgically implanted devices which restore the ability to hear to the hearing impaired. While remarkably successful, even in the best of performers restoration of hearing to levels of normal listeners is unusual. Approximately 3 weeks after surgery, cochlear implants are activated via mapping - a process in which each individual electrode (FDA approved cochlear implants have between 12 and 22 electrodes) is turned on and the stimulus level adjusted to a level that is comfortable and beneficial to the recipient. At present, this standard of care mapping procedure is performed without knowledge of the physical location between the cochlear implant electrodes and the neural interface. Our team has developed a new method of mapping using post-operative CT scans and image processing to specify the physical relationship between the cochlear implant electrodes and the neural interface allowing customized mapping. Using this information, the investigators deactivate sub-optimally positioned electrodes. The investigators term this "Image-guided Cochlear Implant Programming" (IGCIP). In a prospective fashion, the investigators have implemented IGCIP on cochlear implant recipients who have had at least 6 months of standard of care (SOC) mapping. The purpose of this study is to perform a randomized controlled trial (RCT) on newly activated cochlear implant recipients randomizing between IGCIP and SOC.

DETAILED DESCRIPTION:
Over 320,000 individuals have received cochlear implants (CIs) to restore hearing to the hearing impaired. Commercially available CIs have 12, 16, or 22 independent electrodes (the # is dependent on the manufacturer of the CI) which cover the entire frequency spectrum of the cochlea from 20,000 Hertz (Hz) at the base of to 200Hz at the apex. After implantation, an audiologists individually adjusts stimulation levels of each electrode following which all electrodes are turned on such that the whole frequency spectrum of speech can be appreciated. This is known as "standard of care" (SOC) programming. While postoperative speech understanding is significantly better than preoperative levels, even the best performers complain that the fidelity of natural hearing is not reproduced. Additionally, a significant minority achieves poor outcomes despite normally functioning equipment for reasons that are unknown but likely relate to poor neural survival; however, this cannot be confirmed as post-mortem histopathology is required to accurately document spiral ganglion cell count.

In recent years much attention has focused on the interface between the cochlear implant electrodes and the auditory neurons they are stimulating. Technological improvements at Vanderbilt in imaging processing have made it possible to determine the location of each electrode array in relationship to the frequency spectrum of the cochlea.

Using this information, the investigators have developed a new method of CI programming which they call image-guided cochlear implant programming, or IGCIP in which sub-optimally placed electrodes are turned-off or deactivated. Sub-optimally placed electrodes are defined as ones for which their neighboring electrodes are in closer proximity to the site of their neural stimulation. By deactivating sub-optimally positioned electrodes, channel interaction is reduced allowing a cleaner signal to be presented to the auditory nerve.

The investigators have implemented this strategy on 133 CIs of post-lingually deafened (hearing loss after the ability to speak) adult CI users with median use of their CI's with SOC programming of 1.3 years (range 0.3-15.5). When trialing IGCIP, mean word scores increased from 48.8±23.7% to 53.3±22.8% correct, and mean sentence scores increased from 62.2±28.5% to 65.0±26.9% correct. Both of these finding were statistically significant. Extracting out the pre-lingually (hearing loss before the ability to speak) deafened adults, the investigators see that for word scores, 24 of the 133 (28%) had statistically significant improvement 12 of the 133 (9%) had statistically significant decline, and the remaining 97 (73%) had equivocal results. Similarly, for the sentence scores, 36 of the 133 (27%) had statistically significant improvement 24 of the 133 (18%) had statistically significant decline, and the remaining 73 (55%) had equivocal results.

Perhaps the most important metric is which map patients select for long term use - SOC or IGCIP. Ninety-six of the 133 (72.1%) participants elected to keep IGCIP for long term use despite prior research that shows that there is a bias for CI recipients to favor their original map over a new map. And, for the 28% for elected to keep their SOC map, the process involves no risk - the deactivated electrodes are simply reactivated. Given these exciting prospective findings, the investigators are now proposing a randomized controlled trial (RCT) for newly activated adult CI recipients with both the CI user and testing audiologist blinded as to program (SOC or IGCIP). The investigators hypothesize that CI recipients randomized to IGCIP will have improved hearing performance as assessed by both word and sentence testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age that have undergone diagnostic testing for sensorineural hearing loss and are candidates for cochlear implantation will be considered eligible for the study

Exclusion criteria:

* Age < 18 years
* Pre-lingual onset of deafness
* Mini-Mental State Exam < 24 (to remove cognitive decline as a confounding variable)
* Congenital inner ear malformation as detected on pre-operative CT scan performed as routine care
* Non-English speaking (because our audiological speech testing battery is validated for English speakers)
* Have undergone cochlear implantation outside of the Vanderbilt system
* Pregnancy which is a contraindication for elective CT scanning and surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
AzBio Sentence Scores at +5 Signal to Noise Ratio (SNR) | Month 1 post cochlear implant activation
AzBio Sentence Scores at +5 Signal to Noise Ratio (SNR) | Month 3 post cochlear implant activation
AzBio Sentence Scores at +5 Signal to Noise Ratio (SNR) | Month 6 post cochlear implant activation

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Labadie, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Benoit M. Dawant, PhD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No